CLINICAL TRIAL: NCT00828555
Title: Effectiveness of a Vaccination Program in the Community Ob/Gyn Setting
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00011038
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-09

CONDITIONS: Influenza Vaccine; Papillomavirus Infection; Pertussis
Keywords: HPV vaccine; Tdap vaccine
MeSH Terms: conditions — Influenza, Human; Papillomavirus Infections; Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Vaccination Program — Design & implement a program for Ob/Gyns to vaccinate women against human papillomavirus, influenza, & pertussis

SUMMARY:
PURPOSE To develop, implement, and evaluate the effectiveness of a program designed to assist community Ob/Gyns in vaccinating adolescent and adult women against vaccine-preventable diseases.

SPECIFIC AIMS

1. Determine the feasibility of implementing a successful vaccination program for adolescent and adult women in Ob/Gyn offices by direct assessment of medical personnel & office staff on their:

   * Attitudes towards vaccination of women against preventable diseases
   * Perceived barriers to implementing a program to vaccinate women in their offices
   * Ideas on how to overcome barriers to successful program implementation
   * Current vaccination practices and office-specific administrative processes
2. Design & implement a program for Ob/Gyns to vaccinate women against human papillomavirus, influenza, & pertussis
3. Determine the effectiveness of the vaccination program based on

   * Pre- and post-program vaccination rates
   * Program satisfaction amongst Ob/Gyn providers and office staff
   * Willingness to continue and possibly extend the program to additional vaccines
4. Quantify the level of support and resources needed to develop and implement the vaccination program

ELIGIBILITY:
Inclusion Criteria:

* 4-5 community Ob/Gyn practices

Ages: 12 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Population Groups:
  Adults
  Minors
  Patients
  Pregnant Women
  Fetuses
Sampling Method: Non-Probability Sample
Enrollment: 3988 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Implementation and measurement of a health services intervention in community or private Ob/Gyn practices to improve the delivery of standard clinical care to vaccinate women against human papillomavirus, influenza, & pertussis. | Full-scale program implementation will cover a 12 month period, tentatively planned to begin in April 2009.

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Swamy, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Westside OBGYN, Burlington, North Carolina
  - DWHA, Durham, North Carolina
  - Atrium OBGYN, Raleigh, North Carolina
  - Blue Ridge OBGYN, Raleigh, North Carolina